CLINICAL TRIAL: NCT01644214
Title: Extended Pessary Interval for Care (EPIC Study): Patient Preference for 3 Verus 6 Month Follow-up
Brief Title: Extended Pessary Interval for Care (EPIC Study)
Acronym: EPIC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Unity Health Toronto (Other)
Collaborators: Women's College Hospital (Other); Mount Sinai Hospital, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PessaryProtocol
Record Dates: First submitted 2012-06-27; First posted 2012-07-19 (Estimated); Last update posted 2019-12-04 (Actual); Status verified 2019-12

CONDITIONS: Pelvic Organ Prolapse; Pessary
Keywords: Pelvic organ prolapse; Pessary
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pessary Check at 3 months (No Intervention): Patients seen at 3 month intervals for pessary check-ups is the most common interval check in our clinic so this arm is considered the control group.
- 6 month Pessary Check (Experimental): Those that will be seen at 6 month follow-up visits for pessary maintenance will be considered the experimental group of the study.
  Interventions: Other: 6 month follow up for pessary check in the clinic setting

INTERVENTIONS:
Other: 6 month follow up for pessary check in the clinic setting — The standard of care is considered to be pessary checks every 3 months, therefore those that are checked every 6 months will be considered to be in the intervention group.
  Arms: 6 month Pessary Check

SUMMARY:
Objectives: Pelvic organ prolapse (POP) is a common condition for which pessaries are commonly used in conservative treatment. Despite their prevalence, there is no literature to guide the management of pessaries. Our objective is to determine whether patients managed with a pessary for POP are more satisfied with follow-up at 3 or 6 month intervals and if there is any difference in complications rates between the two groups.

Hypothesis: The investigators hypothesize that there will be higher patient satisfaction in the group randomized to 6 month follow-up intervals and that there will be no difference in complication rates between the two follow-up groups.

Method: The investigators will conduct a prospective randomized control trial comparing patient satisfaction and complication rates between patients with pessaries randomized to either 3 or 6 month follow-up intervals over 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Females with POP who have opted for conservative management with a pessary
* Able to read and write English
* First time pessary users
* Successful fitting with a covered ring or Gellhorn pessary, as determined at the usual early follow-up visit 2-4 weeks after initial fitting (successful defined as: no expulsion on movement, squatting or valsalva, no urinary retention, no discomfort, and still retained pessary after 2 weeks)
* Patients agree to use vaginal estrogen (either tablet or cream twice weekly) during the study period; patients may not use a vaginal estrogen ring since this requires changing every 3 months, and will interfere with the study follow-up schedule

Exclusion criteria:

* Current presence of vaginal bleeding, vaginal abrasions or ulcers, or vaginal infection
* Significant cognitive impairment
* Pessary used for indication other than POP (ie. urinary incontinence)
* Use of a pessary that is not a covered ring or Gellhorn (i.e exclude cube, donut, etc.)
* Contraindications to vaginal estrogen
* Unsuccessful pessary fitting (successful defined as: no expulsion on movement, squatting or valsalva, no urinary retention, no discomfort, and still retained pessary after 2 weeks)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2016-11; Primary Completion 2019-11 (Actual); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction | At 6 months from study enrollment
  To determine if patients managed with a pessary for POP are more satisfied with follow-up at 6 or 12 weeks over a one year period.
Patient satisfaction | At 12 months from study enrollment
  To determine if patients managed with a pessary for POP are more satisfied with follow-up at 6 or 12 weeks over a one year period.

SECONDARY OUTCOMES:
Pessary associated complications | Checked at all follow-up visits (3 and 6 months, depending on study group)
  To determine if there is a difference in complication rates associated with indwelling pessaries between those that are seen at 6 week intervals and those that are seen at 12 week intervals, over a one year time period.

CONTACTS AND LOCATIONS:
Overall Officials: Colleen D McDermott, MD, FRCSC, Principal Investigator — St. Michael's Hospital, Women's College Hospital, University of Toronto
Locations (1):
- Women's College Hospital/Mount Sinai Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Samuelsson EC, Victor FT, Tibblin G, Svardsudd KF. Signs of genital prolapse in a Swedish population of women 20 to 59 years of age and possible related factors. Am J Obstet Gynecol. 1999 Feb;180(2 Pt 1):299-305. doi: 10.1016/s0002-9378(99)70203-6. PMID 9988790
- [Background] MacLennan AH, Taylor AW, Wilson DH, Wilson D. The prevalence of pelvic floor disorders and their relationship to gender, age, parity and mode of delivery. BJOG. 2000 Dec;107(12):1460-70. doi: 10.1111/j.1471-0528.2000.tb11669.x. PMID 11192101
- [Background] Fernando RJ, Thakar R, Sultan AH, Shah SM, Jones PW. Effect of vaginal pessaries on symptoms associated with pelvic organ prolapse. Obstet Gynecol. 2006 Jul;108(1):93-9. doi: 10.1097/01.AOG.0000222903.38684.cc. PMID 16816061
- [Background] Schaffer JI, Wai CY, Boreham MK. Etiology of pelvic organ prolapse. Clin Obstet Gynecol. 2005 Sep;48(3):639-47. doi: 10.1097/01.grf.0000170428.45819.4e. No abstract available. PMID 16012231
- [Background] Atnip SD. Pessary use and management for pelvic organ prolapse. Obstet Gynecol Clin North Am. 2009 Sep;36(3):541-63. doi: 10.1016/j.ogc.2009.08.010. PMID 19932415
- [Background] Pott-Grinstein E, Newcomer JR. Gynecologists' patterns of prescribing pessaries. J Reprod Med. 2001 Mar;46(3):205-8. PMID 11304859
- [Background] Thakar R, Stanton S. Management of genital prolapse. BMJ. 2002 May 25;324(7348):1258-62. doi: 10.1136/bmj.324.7348.1258. No abstract available. PMID 12028982
- [Background] Sarma S, Ying T, Moore KH. Long-term vaginal ring pessary use: discontinuation rates and adverse events. BJOG. 2009 Dec;116(13):1715-21. doi: 10.1111/j.1471-0528.2009.02380.x. PMID 19906018
- [Background] Powers K, Grigorescu B, Lazarou G, Greston WM, Weber T. Neglected pessary causing a rectovaginal fistula: a case report. J Reprod Med. 2008 Mar;53(3):235-7. PMID 18441734
- [Background] Ko PC, Lo TS, Tseng LH, Lin YH, Liang CC, Lee SJ. Use of a pessary in treatment of pelvic organ prolapse: quality of life, compliance, and failure at 1-year follow-up. J Minim Invasive Gynecol. 2011 Jan-Feb;18(1):68-74. doi: 10.1016/j.jmig.2010.09.006. PMID 21195956
- [Background] Lamers BH, Broekman BM, Milani AL. Pessary treatment for pelvic organ prolapse and health-related quality of life: a review. Int Urogynecol J. 2011 Jun;22(6):637-44. doi: 10.1007/s00192-011-1390-7. Epub 2011 Apr 7. PMID 21472447
- [Background] Wu V, Farrell SA, Baskett TF, Flowerdew G. A simplified protocol for pessary management. Obstet Gynecol. 1997 Dec;90(6):990-4. doi: 10.1016/s0029-7844(97)00481-x. PMID 9397117
- [Background] Gorti M, Hudelist G, Simons A. Evaluation of vaginal pessary management: a UK-based survey. J Obstet Gynaecol. 2009 Feb;29(2):129-31. doi: 10.1080/01443610902719813. PMID 19274547
- [Background] Adams E, Thomson A, Maher C, Hagen S. Mechanical devices for pelvic organ prolapse in women. Cochrane Database Syst Rev. 2004;(2):CD004010. doi: 10.1002/14651858.CD004010.pub2. PMID 15106231
- [Background] Crandall C. Vaginal estrogen preparations: a review of safety and efficacy for vaginal atrophy. J Womens Health (Larchmt). 2002 Dec;11(10):857-77. doi: 10.1089/154099902762203704. PMID 12626086
- [Derived] Bugge C, Adams EJ, Gopinath D, Stewart F, Dembinsky M, Sobiesuo P, Kearney R. Pessaries (mechanical devices) for managing pelvic organ prolapse in women. Cochrane Database Syst Rev. 2020 Nov 18;11(11):CD004010. doi: 10.1002/14651858.CD004010.pub4. PMID 33207004